CLINICAL TRIAL: NCT00722709
Title: Randomised Double Blind Trial to Investigate the Effects of Intraperitoneal Local Anaesthetic Following Colonic Surgery.
Brief Title: Intraperitoneal Local Anaesthetic in Colonic Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Dr Arman Kahokehr, University of Auckland
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAstudy
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Colon Surgery
Keywords: Pain; Fatigue; Colon; Surgery; ERAS; Fastrack; Local anaesthetic; Peritoneum; Metabolic; Endocrine; Post surgical metabolic response; Complications; Time to passage of flatus; Time to passage of stool; Time to discharge from facility; Re-admission rate
MeSH Terms: conditions — Pain; Fatigue | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LA (Experimental): Use of Ropivacaine
  Interventions: Drug: Ropivacaine
- Placebo (Placebo Comparator): Use of 0.9% saline
  Interventions: Drug: 0.9% Saline

INTERVENTIONS:
Drug: Ropivacaine — In the treatment arm patients will receive 10mls 0.75% ropivacaine diluted to 50mls with saline immediately before closure.
  At closure, two small 2 mm catheters will be placed in the peritoneal cavity at the site of the operation to infuse local anaesthesia. This will penetrate through the skin once closure is complete. This will be attached to a small infusion pump (On-Q pain buster). This pump will contain 270mls of 0.2% ropivacaine. After 68 hours the pump will be stopped and the catheter will be removed in a similar fashion as routine drain removal.
  Arms: LA
Drug: 0.9% Saline — In the placebo arm patients will receive 50 ml 0.9% saline into the peritoneum soon after the creation of the laparotomy.
  At closure, two 2 mm catheters will be placed in the peritoneal cavity at the site of the operation to infuse local anaesthesia. This will penetrate through the skin once closure is complete. This will be attached to a small infusion pump on-Q pain buster). This pump will contain 0.9% saline. After 68 hours the pump will be stopped and the catheter will be removed in a similar fashion as routine drain removal.
  Arms: Placebo

SUMMARY:
Aim:

The general aim of this research group is to improve the recovery of patients after abdominal surgery. The specific aim of this study is to conduct a randomized, double blinded, controlled trial to investigate the effect of intra-peritoneal local anaesthesia application on postoperative pain and post-operative fatigue. This will be conducted in the setting of an enhanced recovery after surgery program (ERAS).

Methods:

Patients will be randomised by computer generated random numbers and opaque envelope method. In the treatment arm patients will receive 10ml 0.75% ropivacaine diluted to 50mls with 0.9% saline soon after the creation of the laparotomy . In the placebo arm, 50mls of 0.9% normal saline will be used in a similar fashion. At closure, two small 2mm catheter belonging to the On-Q pain buster system will be placed in the peritoneal cavity. This will be attached to a pump which will contain either a 0.2% ropivacaine solution or 0.9% saline placebo running at 4mls/hr for 68 hours. All members involved in patient care (with the exception of one nurse) will be blinded to the above. After 68 hours the pump will be stopped and the catheter will be removed. Assessment of postoperative pain will be performed by visual analogue scale, and fatigue assessment will be done using the Identity Consequence Fatigue Scale (ICFS) at various intervals post-operatively. Blood tests for inflammatory markers including glucose, cortisol, CRP, albumin and several cytokines as well as local anaesthetic levels will be taken.

Significance to health:

This method of analgesia administration has not been investigated in open major colonic surgery. This trial has wide reaching implications, with the potential to improve pain and thus recovery after abdominal surgery.

DETAILED DESCRIPTION:
Scientific Background:

Postoperative fatigue (POF) is a common phenomenon following abdominal surgery and is currently under investigation at the department of surgery, Middlemore hospital, Auckland. POF in patients undergoing major abdominal procedures is very common. It has been reported that 92% of patients who have undergone abdominal surgery report increased fatigue reports immediately after the procedure, dropping to about 10% in 3 months. POF comprises of unpleasant symptoms that impact on the patient's quality of life.

1. It can create difficulties in performing activities of daily living.
2. The symptoms of POF include tiredness, lack of energy and sense of debilitating muscle weakness.
3. POF is thought to be associated with poor physical, psychological and functional outcomes.
4. The aetiology of POF is thought to be multi-factorial. Biological, psychological and social factors all contribute.

The biological aspect of POF can be divided into the physiological stress response to the trauma of surgery, postoperative nutritional deficits and the loss of previous cardiovascular fitness subsequently after surgery. Various methods have been investigated over the last two decades to address and "dampen" the physiological response in order to enhance postoperative recovery.

There are two possible ways of communication between the periphery and the brain. One is the hormonal route and the other is the neural route. The later route is projected via paracrine action of local cytokines on the afferent nerve endings 5. In the abdominal cavity, there are two types of afferent endings 6. These are the vagal afferents and spinal afferents. Vagal and spinal afferent fibres transmit sensory information from the GI tract to the CNS. Afferents from the vagus nerve conduct neuronal messages from the intra-peritoneal cavity to the CNS.

Vagal afferents have cell bodies in nodose ganglia and enter via the brainstem. In comparison cell bodies of the spinal afferents are located in the dorsal root ganglion and project to the dorsal horn of the cord. They follow the paths of the sympathetic and parasympathetic efferents to the gut wall.

Vagal afferents are either intramuscular or intraganglionic. Spinal afferents on the other hand are located in the serosa, mesenteric attachments and the submucosa of the tract.

The surgical stress response produces alterations in the haemodynamic, metabolic and immune response of patients 7. The biochemical cytokine response to surgical trauma is well understood and summarised well by Ni Choileain.

There are elements of immune over stimulation resulting in a cascade of cytokine activation following surgery. These cytokines include tumour necrosis factor alpha (TNF-a) and interleukin 1B (IL-1B). These can stimulate the production and release of other cytokines including interleukin 6 (IL-6). IL-6 results in the production of C-reactive protein (CRP) and other acute phase proteins through the hepatic component of this response.

Therapeutic strategies are aimed at restoring these physiological imbalances associated with surgery.

In the rat sub diaphragmatic vagotomy has prevented the effects of intraperitoneal IL-1 administration which prevented increases in body temperature and the increase in secreted hypothalamic norepinephrine (NE), and markedly attenuated the increases in plasma ACTH and corticosterone 8. This is thought to have reduced the "sickness response" to intraperitoneal cytokine administration. Similarly, administration of localised partial body exposure to irradiation in vagotomised rats resulted in decreased hypothalamic, thalamic, hippocampal and cortical IL-6, IL-1b and TNF-a compared with non-vagotomised rats 9. It is therefore thought that the vagus plays a major role in the surgical stress response although it is important to point that the vagus is not thought to be solely responsible for the activation of hypothalamic activity 10.

A pro-inflammatory cytokine pathway after abdominal surgery, with direct action of cytokines on the vagus nerve as a major vehicle in this response, is therefore, a feasible explanation for contributing to POF.

In the clinical context, recent developments in elective large bowel surgery include the use of Fast Track (FT) or Enhanced Recovery After Surgery (ERAS) protocols. The use of such protocols is generally said to affect metabolic, neural and other organ activities in order to reduce morbidity, increase recovery time and result in shorter hospital stays.

There are numerous elements to these protocols, given there are multiple contributors to POF, as already discussed. In brief, some of these interventions include extensive preoperative counseling and preparation psychologically, no preoperative fasting, carbohydrate loading, use of epidural anaesthesia, avoidance of peri-operative fluid over load, early removal of catheters, drains and early mobilisation with physiotherapist. 11.

Other interventions, such as pre-operative steroid administration, are currently being trialed as part of an ERAS surgical protocol at the Manukau Surgery Centre (MSC), Middlemore Hospital, Auckland. The purpose is to enhance recovery by decreasing the cascade of pro-inflammatory post surgical response using the immunosuppressive properties of this agent. As discussed earlier, pro-inflammatory responses are hypothesised to contribute to POF.

Local anaesthetic (LA) agents, when applied in sufficient concentration at the site of action, prevent conduction of electrical impulses by the membranes of nerve and muscle12. In order to obtain a clear picture of the fundamental blocking mechanism, knowledge of the channel-binding kinetics of the drug is necessary. The application of LA agents to the intraperitoneal cavity has been investigated in several trials to decrease post operative pain and enhance recovery 13-18. Unfortunately there are few studies if any looking at the application of local anaesthesia in open procedures compared with laparoscopic gastrointestinal procedures. It is therefore an area where trials are needed.

It is not unreasonable that the application of local anaesthesia to the intraperitoneal cavity should play a role in ERAS protocols. In order to reduce postoperative pain and reduce intra-abdominal to CNS signal transmission we will produce a transient "chemical affarenectomy". As part of the already established ERAS protocol at the Manukau Surgical Centre (MSC), my aim is to look at the effects of instillation of local anaesthesia to the intra-peritoneal cavity immediately after opening the abdominal cavity and we propose an ongoing LA infusion with an intraperitoneal catheter and external pump postoperatively.

Objectives:

1. To be involved in running the already established ERAS program at Manukau Surgical Centre (MSC).
2. Conduct a randomised double blinded controlled trial to investigate the effect of intra-peritoneal local anaesthesia application on postoperative pain and POF in patients under the ERAS protocol.

Methods and Outcomes:

There is already an established ERAS perioperative care plan at the MSC. Patients are usually recruited from surgical outpatients clinics at Manukau Super Clinic. Patients who are undergoing colonic operations are recruited in the ERAS program under the supervision of the primary consultant colorectal surgeon. My aim is to be involved in data gathering and clinical aspects of maintaining this protocol.

Summary of ERAS perioperative care plan at MSC conducted by Zargar et al. (Table 1)

* Pre-Operative Information and counseling
* Carbohydrate Loading
* Avoidance of Mechanical Bowel Preparation
* Continuous Bupivacaine thoracic epidural analgesia
* Limited IV fluid therapy (ERAS anaesthetic protocol)
* Avoidance of prophylactic nasogastric tubes
* Early Post operative oral intake
* Dietary Supplementation
* Avoidance of opioids
* Early mobilisation according to mobilisation protocols
* Discharge Criteria

Research Design:

Randomised double blinded clinical trial to investigate the effects of washing and infusing the intraperitoneal cavity with local anaesthesia on postoperative pain and fatigue scores on patients undergoing open colonic procedures.

Ethics:

Ethics approval for this project has been obtained.

Sample size:

Using the data from a previous study in measuring post-operative fatigue following colonic surgery, in order to detect a reduction of post-operative fatigue by 30% on day 7 post-operatively with alpha of 0.05 and power of 0.8, 21 patients are required in each group, we will aim for 30 patients in each arm anticipating for possible drop outs.

Brief Method:

Patients will be randomised by computer generated random numbers and opaque envelope method. In the treatment arm patients will receive 10mls 0.75% ropivacaine diluted to 50mls with 0.9% saline soon after the creation of the laparotomy or in the placebo arm, receive 50mls of 0.9% normal saline in a similar fashion. One theatre staff nurse who will not be involved in patient care will be given the blinded envelop and prepare the lidocaine or saline mixtures in the theatre drug room. The mixtures will be unlabelled and appear similar in color. These will be given to the surgeon during the procedure. All members of the staff involved in patient care including the anaesthetist will be blinded to the solution administered.

The theatre staff nurse will then prepare a small infusion pump. The mixture used in the pump will be pre-mixed by one of the clinical pharmacists at Middlemore hospital who will not be involved in patient care. The staff nurse will be un-blinded to the contents of the mixtures. The nurse will prepare the pump and load either the anaesthetic or saline solution. At closure, two small 2mm catheter will be placed in the peritoneal cavity at the site of the operation to infuse local anaesthetic. This will penetrate through the skin once closure is complete. This will be attached to a small infusion pump (On-Q pain buster). This pump will contain either a 270mls of 0.2% ropivacaine or 270mls of 0.9% saline. All members involved in patient care including surgical, anaesthetic and nursing teams will be blinded to the contents of this pump. The pump will be activated at a set rate of 4mls/hr immediately once the patient is in the post anaesthesia recovery room. The pump will run continuously. The patient will continue recovery on the ward as per ERAS protocol. After 68 hrs the pump will be stopped and the catheter will be removed in a similar fashion as routine drain removal.

Endpoints:

* Assessment of postoperative pain using Visual analogue scale (VAS) 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, day 1, day 2 and day 3 post operatively.
* Forced expiratory volumes using a peak flow meter immediately pre-operatively in the anaesthesia room and 1 hour, 2 hours, 4 hours, 8 hours, day 1, day 2 and day 3 postoperatively (best of 3 attempts for each measurement will be used)
* Fatigue assessment will be done using the Identity Consequence Fatigue Scale (ICFS) pre-operatively and on day 1, 2 and 3, 7, 30 and 60 postoperatively respectively.
* Serum Glucose, cytokines and local anaesthetic level at 8, 20, 48, 72 hours post op.
* CRP, Albumin at 20, 48 and 72 hours post op.

Resources:

Consultant Colorectal Surgeons at Middlemore Hospital involved in the project: Associate Professor Andrew Hill, Mr Andrew Connolly and Mr Lincoln Israel.

Consultant anaesthetist:

Matthew Taylor Patients- approximately 100 major colorectal resections are performed at MSC per year.

Manukau Surgical Centre staff facilities University of Auckland facilities

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients undergoing open colonic resection at MSC under the ERAS program.

Exclusion Criteria:

* Known sensitivity to the local anaesthetic agents
* Patients who prefer not to participate (no consent gained)
* ASA greater or equal to 4
* Rectal resection
* Formation of stoma
* Current use of systemic steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-11 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Post operative recovery using the Identity consequence fatigue scale (ICFS) | Base-line, Day 1, Day 3, Day 7, Day 14, Day 30, Day 60

SECONDARY OUTCOMES:
Post-operative rest, movement and cough pain using Visual analogue score | 2,4,6,8,12,24,48,72 hours and on day 7
Post operative analgesia use using morphine equivalence data | Total use on day 1, day 2, day 3 post operatively and total use until discharge
Serum Ropivacaine level, serum Cytokine, serum Cortisol, serum glucose and serum CRP. Albumin, haematological parameters and biochemical parameters. | Pre-operatively, 8, 20, 48,72 hours post operatively
Questions aimed at symptoms of local anaesthetic toxicity | 2, 4, 6, 8, 12, 24, 48, 72 hours post operatively
Recovery of bowel function measured by time to pass flatus and time to pass stool post-operatively. | Assessed at 2, 4, 6, 8, 12, 24, 36, 48, 60, 72 hours.
Quality of care assessment based on a 100mm visual analogue scale (1-10). | pre-op, day1, day 2, day3, day 7, day 30 and day 60 post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Arman A Kahokehr, MBChB, Study Director — University of Auckland, New Zealand; Andrew G Hill, FRACS, Principal Investigator — University of Auckland, New Zealand
Locations (2):
- New Zealand (2):
  - Manukau Surgery Centre-Middlemore Hospital, Auckland, Auckland
  - University of Auckland, Auckland, Auckland

REFERENCES:
- [Derived] MacFater WS, Xia W, Barazanchi AWH, MacFater HS, Lightfoot N, Svirskis D, Kahokehr AA, Hill AG. Association between perioperative intraperitoneal local anaesthetic infusion and long-term survival and cancer recurrence after colectomy: follow-up analysis of a previous randomized controlled trial. ANZ J Surg. 2020 May;90(5):802-806. doi: 10.1111/ans.15753. Epub 2020 Feb 23. PMID 32090464
- [Derived] Kahokehr A, Sammour T, Zargar Shoshtari K, Taylor M, Hill AG. Intraperitoneal local anesthetic improves recovery after colon resection: a double-blinded randomized controlled trial. Ann Surg. 2011 Jul;254(1):28-38. doi: 10.1097/SLA.0b013e318221f0cf. PMID 21670611